CLINICAL TRIAL: NCT01753700
Title: Effect of UHT Treated Milk on Blolipid Profile
Acronym: UHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Arla Foods (Industry); Hoeng Fonden (Unknown); Bionor Pharma (Unknown)
Responsible Party: Principal Investigator, AAstrup, MD, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B300
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: To Investigate the Effect of UHT Treated Milk Versus Pasteurised Milk on Bloodlipid Profil
Keywords: crossover; UHT milk; Pasteurised milk; supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UHT treated milk (Experimental): 1,5 L of 1,5% UHT milk pr day for 3 weeks (21days)
  Interventions: Dietary Supplement: UHT treated milk
- Paseurised milk (Placebo Comparator): 1,5 L 1,5% pasteurised milk pr day for 3 weeks (21 days)
  Interventions: Dietary Supplement: UHT treated milk

INTERVENTIONS:
Dietary Supplement: UHT treated milk

SUMMARY:
The studie are to investigate the effect of ultra heat treated (UHT) versus pasteurised milk on bloodlipid profile

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* 22-50 years of age
* BMI 25-30
* non smokers

Exclusion Criteria:

* lactose intolerance
* milk allergy or other types of food allergy
* Intestinal, abdominal or endocrinnologic diseases
* daily use of dietary supplements incl. vitamins and minerals
* cronic diseases (diabetes, CVD etc.)
* user of medicin on perscription that can influence the resuts of the study
* allergic to paraamino benzoe acid
* Physical activity > 10 h pr week
* Blood donor
* on a diet or change of dietary habits within 3 months
* body weigh change > 3 kg within the last 3 month
* special diets
* concomitant participation on other studies
* not able to comply with protocol

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Blood lipids | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Frederiksberg, Denmark